CLINICAL TRIAL: NCT04355715
Title: Evaluation of a COVID-19 Screening Strategy Combining Chest Low Dose CT and RT-PCR Test for Patients Admitted for Surgical or Interventional Procedures During the COVID 19 Outbreak
Brief Title: Combination of Chest Scanography and Nasal Viral Detection Test to Detect COVID-19 Positive Patients Before Surgical Intervention in a University Hospital During Coronavirus Pandemia
Acronym: COVID-Scan
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0223
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID 19; SARS-Cov-2
Keywords: COVID-19 infection or paucy-symptomatic carriage; In-hospital screening; Chest CT-scan
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Plasma: preoperative, ICU admission at POD0 and POD1 samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to improve the screening for COVID-19 upon admission to the Montpellier University Hospital for an act under general anesthesia or at high risk of transmission of the virus. Indeed, routine nasal swabs present many false negatives (60 to 70%) and many patients with the coronavirus have little or no symptoms. Performing a chest CT scan can reveal early signs very suggestive of viral pneumoniae due to the new coronavirus without additional risk compared to a simple chest X-ray (no injection of contrast medium, low exposure).

The objective is to assess the sensitivity of the diagnosis of COVID-19 by carrying out a nasopharyngeal RT-PCR and a low dose thoracic scanography at the hospital admission of patients scheduled to a procedure under general anesthesia or at risk of aerosolization (surgery, endoscopy, procedures involving risk of interventional radiology) in order to limit the risks of transmission to healthcare professionals or other patients and to rationalize the use of protective equipment.

This is an observational research without modification of care in the setting of COVID-19 pandemia. All clinical and biological data will be issued from routine care and medical charts. Routine use of CT scan and nasal swabs is an institutional approved strategy. Serologic tests will be performed as soon as available from serum collection collected after routine blood analysis. All data will be anonymously recorded after information and non-opposition of the patient.

ELIGIBILITY:
Inclusion criteria:

* Scheduled or unscheduled surgical or interventional procedure with at least one night in hospital
* Chest CT-scan within the first 24 hours
* Nasopharyngeal swaps within 24 hours before or after hospital admission

Exclusion criteria :

* Age under 18 years
* Patient with restriction of freedom
* Vital surgical emergency
* Direct admission to the COVID dedicated hospital
* Opposition to data utilization

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital for a surgical or interventional procedure under general anesthesia or at risk of aerosolization during the COVID-19 outbreak and screened with chest CT-scan and nasopharyngeal RT-PCR to detect SARS-Cov-2 infection or carriage
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Confirmed diagnosis of COVID-19 infection | 15 days
  One of the following criteria: Viral pneumonia, positive COVID-19 RT-PCR, or COVID-19 seroconversion (new onset of specific IgM or increased rate of specific IgG)

SECONDARY OUTCOMES:
Incidence of unexpected COVID-19 positive patients admitted to the hospital | 24 hours from hospital admission
  Number of patients admitted to the hospital for an invasive procedure with COVID-19 detected by the combined strategy CT-scan plus RT-PCR at admission
Number of contaminating events avoided by the early detection of COVID-19 patients | Hospital stay up to 15 days
  Number of events at high risk of viral transmission performed under accurate protection in COVID-19 patients detected by the early combined strategy, among hospitalization, unprotected in-hospital transportation, unprotected invasive procedure, in-bed chest X-ray, respiratory physiotherapy.
Incidence of SARS-Cov-2 seroconversion | 15 days
  Modification of serologic status between hospital admission and day 15 or hospital discharge which ever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gaudard, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC